CLINICAL TRIAL: NCT02117518
Title: Selective Immunotargeting of Pathogenic CD8 T Cells of Type 1 Diabetes Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Migal Galilee Research Institute (Other)
Collaborators: Ziv Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0063-13
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Type I Diabetes
Keywords: type 1 diabetes; autoreactive T cells; beta cell peptides; genetically modified T cells; mRNA electroporation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: T1D patients at ages 0-25
  Interventions: Other: blood drawing

INTERVENTIONS:
Other: blood drawing

SUMMARY:
It is well established that CD8 and CD4 T cells reactive against defined islet antigens are associated with initiation and progression of Type 1 Diabetes (T1D). In previous work, we have demonstrated that it is possible to redirect T cells against pathogenic T cells via chimeric peptide/MHC/CD3-zeta receptors in a peptide-specific manner and to prevent, or inhibit diabetes in NOD mice. In this study we intend to extend this approach to T cells of T1D patients. Working hypothesis: Beta cell-reactive CD8 T cells of human T1D patients can be immuno-targeted by their own gene-modified cytotoxic T lymphocytes (CTLs). Aims: Our major aim is to demonstrate, in a set of ex-vivo experiments, such immunotargeting with T cells derived from T1D patients at the Ziv Medical Center. To this end we will stimulate and expand autoreactive CD8 cells in blood samples of T1D patients and target them, ex-vivo, with genetically-reprogrammed CTLs which are present in the same blood samples.

DETAILED DESCRIPTION:
To obtain proof-of-principle of our approach we have initiated tight collaboration between the Laboratory of Immunology at MIGAL Galilee Research Institute, Kiryat Shmona (MIGAL) and Breinin Center for Type 1 Diabetes and Endocrinology at the Ziv Medical Center in Safed (Ziv). In this study we will first identify carriers of the HLA-A0201 allele among pediatric and young adult T1D patients at Ziv. We will then screen the T cell pool in the peripheral blood samples of these patients for CD8 T cells reactive against any of 3 known HLA-A0201-binding peptides associated with autoreactivity in T1D: Insulin beta chain 10-18, IGRP 265-73 and IGRP 222-230. The influenza virus-derived peptide MP 58-66 will serve as reference. Next we will isolate polyclonal CD8 T cells from blood samples of the same patients, activate and expand them ex-vivo and transfect them via electroporation with in-vitro-transcribed mRNA encoding the respective peptide/MHC/CD3-zeta construct(s). We will then perform co-culture experiments assessing the ability of the mRNA-transfected T cells to kill the autoreactive T cells of the same patient in a peptide-selective manner.

ELIGIBILITY:
Inclusion Criteria:

* Children and young adults, ages between 0-25 who were diagnosed with T1D no more than 3 years prior to enrollment.

Exclusion Criteria:

* none

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: T1D patients who were diagnosed up to 3 years prior to recruitment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Identification, isolation, propagation and targeting of autoreactive T cells from T1D patients | 2 years from the final approval of study
  The ability of the genetically-modified cells to target and kill target autologous autoreactive CD8 T cells will be analyzed by CFSE and HLA-I tetramer staining using flow cytometry and IFN gamma production using ELISPOT.

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Gross, PhD, Study Director — Migal Galilee Research Institute; Orna Gottfried, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel